CLINICAL TRIAL: NCT02613286
Title: A Proof of Concept Non-inferiority Trial Evaluating the Safety and Efficacy of Extrafascial Hysterectomy Plus Pelvic Lymph-node Dissection in Patients With Stage IA2-IB1 Cervical Cancer ≤ 2cm
Brief Title: LESs Surgical Radicality for EaRly Stage Cervical Cancer
Acronym: LESSER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Câncer de Pernambuco (Other)
Collaborators: Santa Casa de Misericórdia de Maceió (Other); Professor Fernando Figueira Integral Medicine Institute (Other)
Responsible Party: Principal Investigator, Thales Paulo Batista, Consultant Physician and Researcher (Surgical Oncology), Hospital de Câncer de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAAE: 42981715.7.0000.5205; U1111-1176-6929 (Other: UTN/WHO)
Record Dates: First submitted 2015-11-20; First posted 2015-11-24 (Estimated); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Uterine Cervical Neoplasms
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: Proof of concept design (phase II non-inferiority trial)
Who Masked: Participant
Masking Description: Due to the surgical nature of the study, only participants were masked to treatment allocation
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Extrafascial Hysterectomy (Experimental): Type A hysterectomy with 1 - 2cm of vaginal cuff plus level 1 pelvic lymph-node dissection according to Querleu and Morrow classification.
  Interventions: Procedure: Extrafascial Hysterectomy
- Modified radical hysterectomy (Active Comparator): Type B2 hysterectomy with 1 - 2cm of vaginal cuff plus level 1 pelvic lymph-node dissection according to Querleu and Morrow classification.
  Interventions: Procedure: Modified radical hysterectomy

INTERVENTIONS:
Procedure: Extrafascial Hysterectomy — Hysterectomy plus Pelvic Lymph-Node Dissection
  Arms: Extrafascial Hysterectomy
Procedure: Modified radical hysterectomy — Hysterectomy plus Pelvic Lymph-Node Dissection
  Arms: Modified radical hysterectomy

SUMMARY:
This study is an open-label, multicenter, randomized, phase II non-inferiority trial (proof of concept study). Its purpose is to evaluate the safety and efficacy of extrafascial hysterectomy plus pelvic-lymph node dissection compared with the standard modified radical hysterectomy in patients with stage IA2-IB1 cervical cancer ≤ 2cm.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and efficacy of extrafascial hysterectomy compared with modified radical hysterectomy, both plus level 1 pelvic lymph-node dissection, in patients with early stage IA2-IB1 cervical cancer ≤ 2cm. The experimental procedure will be considered to be promising for treatment of stage IA2-IB1 cervical cancer ≤ 2cm if the Bayesian posterior probability of "the difference of the 3-y DFS rate is less than the non-inferiority margin of 5%" is at least 50%. Thus, using this proof of concept design, the planned sample size is 40, with 20 cases per arm, which provides 72% chance of satisfying the above criteria, under the hypothesis that the lowest 3-y DFS rate in each arm is 90%. As required, adjuvant therapy will include cisplatin-based chemo-radiation or pelvic radiation alone (EBRT +/- intracavitary brachytherapy) indicated according to the #GOG92 and #GOG109 criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed adenocarcinoma, squamous, or adenosquamous cancer of the cervix by LEEP, cone or cervical biopsy;
2. Aged between 18 and 70 years;
3. performance status 0-2 (ECOG, Eastern Cooperative Oncology Group) and / or greater than 70 points by the Karnofsky scale;
4. FIGO early stage IA2-IB1 ≤ 2cm;
5. Appropriated cardio-respiratory, hepato-renal and hematological reserves; and
6. Signing of the Consent Form.

Exclusion Criteria:

1. Limiting systemic comorbidities including neuro-psychiatric disorders or obesity;
2. Apparent or confirmed uncontrolled infections;
3. Other malignancies in activity;
4. Previous radiation or chemotherapy treatment or major pelvic surgery;
5. History of drug allergies, and pregnancy or breast feeding; and
6. Evidence of more extensive disease at the time of surgery.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2022-05-10 (Actual)

PRIMARY OUTCOMES:
Disease Free Survival (3-y DFS) | 3 years
  Time from surgery to recurrence

SECONDARY OUTCOMES:
Treatment-related adverse events (surgical) | 90 days
  Surgical morbidity and mortality
Patient reported QoL | Base-line and 6 months.
  QoL according to EORTC C30 questionnaire (v3.0)
Rates of using adjuvant therapy | 90 days
  Cisplatin-based chemo-radiation or pelvic radiation alone (EBRT +/- intracavitary brachytherapy) indicated according to the #GOG92 and #GOG109 criteria
Overall survival (3-y OS) | 3 years
  Time from surgery to death of any cause

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carneiro VCG, Batista TP, Andrade MR, Barros AV, Camara LHLD, Ramalho NM, Lucena MA, Fontao DFS, Tancredi R, Silva Junior TC, Bezerra ALR, Baiocchi G. Proof-of-concept randomized phase II non-inferiority trial of simple versus type B2 hysterectomy in early-stage cervical cancer </=2 cm (LESSER). Int J Gynecol Cancer. 2023 Apr 3;33(4):498-503. doi: 10.1136/ijgc-2022-004092. PMID 36696980